CLINICAL TRIAL: NCT02056782
Title: A Pilot Study to Evaluate the Safety and Preliminary Evidence of an Effect of ODSH (2 O, 3-O Desulfated Heparin) in Accelerating Platelet Recovery in Patients Receiving Induction or Consolidation Therapy for Acute Myeloid Leukemia
Brief Title: A Pilot Study of Dociparstat Sodium (ODSH) in Acute Myeloid Leukemia
Acronym: PGX-AML
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Collaborators: Translational Drug Development (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PGX-ODSH-2013-AML-1
Record Dates: First submitted 2014-01-22; First posted 2014-02-06 (Estimated); Results first posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2022-05

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; AML; ODSH; ODSH-AML; CX-01; dociparstat; dociparstat sodium; 2-O, 3-O desulfated heparin
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — N-desulfated,2-O,3-O-desulfated heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dociparstat (Experimental): The following induction regimen was administered:
  * Cytarabine (100 mg/m2/day) via continuous intravenous (IV) infusion 24 hours daily for 7 days.
  * Idarubicin (12 mg/m2/day) IV on Days 1, 2, and 3.
  * Dociparstat (4 mg/kg) given over 5 minutes IV, immediately after the idarubicin dose on Day 1, followed by a continuous IV infusion (0.25 mg/kg/hr for 24 hours daily) for a total of 7 days.
  Interventions: Drug: Dociparstat sodium

INTERVENTIONS:
Drug: Dociparstat sodium — The following induction regimen was administered:
  * Cytarabine (100 mg/m2/day) via continuous intravenous (IV) infusion 24 hours daily for 7 days.
  * Idarubicin (12 mg/m2/day) IV on Days 1, 2, and 3.
  * Dociparstat (4 mg/kg) given over 5 minutes IV, immediately after the idarubicin dose on Day 1, followed by a continuous IV infusion (0.25 mg/kg/hr for 24 hours daily) for a total of 7 days.
  Other Names: dociparstat; ODSH; CX-01; 2-O, 3-O desulfated heparin

SUMMARY:
This was an open-label pilot study that evaluated the safety and preliminary evidence of a therapeutic effect of dociparstat in conjunction with standard induction and consolidation therapy for acute myeloid leukemia (AML).

DETAILED DESCRIPTION:
The primary objectives of this study were the following:

1. To evaluate the safety and tolerability of dociparstat in patients with acute myeloid leukemia (AML) receiving cytarabine and idarubicin induction or cytarabine consolidation chemotherapy.
2. To determine whether there is preliminary evidence of an effect of dociparstat on time to transfusion-independent platelet recovery in AML patients receiving cytarabine and idarubicin induction or cytarabine consolidation chemotherapy.

The secondary objectives of this study were the following:

1. To determine whether there is preliminary evidence of an effect of dociparstat on remission rate following cytarabine and idarubicin induction in AML patients.
2. To determine whether there is preliminary evidence of an effect of dociparstat on improving platelet nadir counts in AML patients receiving cytarabine and idarubicin induction or cytarabine consolidation chemotherapy.
3. To determine whether there is preliminary evidence of an effect of dociparstat on decreasing the number of platelet transfusions in AML patients receiving cytarabine and idarubicin induction or cytarabine consolidation chemotherapy.
4. To determine whether there is preliminary evidence of an effect of dociparstat on reducing overall side effects of chemotherapy in AML patients receiving cytarabine and idarubicin induction or cytarabine consolidation chemotherapy.

This study enrolled patients with newly diagnosed, previously untreated AML; subjects with acute promyelocytic leukemia and acute megakaryoblastic leukemia subtypes were excluded.

All patients were to receive standard induction chemotherapy with cytarabine 100 mg/m2/day by continuous intravenous (IV) infusion over 24 hours daily for 7 days (Days 1-7) plus idarubicin 12 mg/m2/day by IV injection daily for 3 days (Days 1-3). For consolidation, patients younger than 60 were to receive cytarabine at a dose of 3 grams/m2 over 3 hours, every 12 hours on days 1, 3, and 5.

Induction cycle: dociparstat 4 mg/kg IV bolus Day 1, 30 minutes after completion of administration of the first dose of idarubicin, then dociparstat 0.25 mg/kg/hour for 24 hours daily by continuous IV infusion Days 1-7.

Consolidation cycle: dociparstat mg/kg IV bolus Day 1 administered 30 minutes after completion of infusion of the first dose of cytarabine then dociparstat 0.25 mg/kg/hour for 24 hours daily by continuous IV infusion Days 1-5

In total, there were 7 days in the induction cycle and 5 days in the consolidation cycles.

ELIGIBILITY:
Inclusion Criteria:

All patients had to meet the following criteria to be eligible for this study:

1. Had newly diagnosed, previously untreated acute myeloid leukemia (AML). Acute promyelocytic leukemia and acute megakaryoblastic leukemia subtypes were excluded
2. Had no prior chemotherapy for AML; however, prior hydroxyurea to control white blood cell count was allowed
3. Was aged 18 years or older.
4. Had an Eastern Cooperative Oncology Group (ECOG) Performance status of 0-2.
5. Had a cardiac ejection fraction ≥ 50% (echocardiography or Multi-Gated Acquisition Scan [MUGA]).
6. Had adequate hepatic and renal function (aspartate aminotransferase [AST], alanine aminotransferase [ALT], bilirubin and creatinine < 2.5 x upper normal limit).
7. Was able to provide informed consent and signed an approved consent form that conformed to federal and institutional guidelines.

Exclusion Criteria:

Patients who met any of the following criteria were not eligible to be enrolled in this study:

1. Had acute promyelocytic leukemia.
2. Had acute megakaryoblastic leukemia.
3. Had central nervous system (CNS) leukemia
4. Had the presence of uncontrolled bleeding.
5. Had the presence of significant active infection that was uncontrolled, as judged by the Investigator.
6. Had a history of severe congestive heart failure or other cardiac disease that contraindicated the use of anthracyclines, including idarubicin.
7. Had pre-existing liver disease.
8. Had renal insufficiency, which, in the opinion of the Investigator, might have adversely affected the schedule and dose of therapy with cytarabine, as well as the management of tumor lysis syndrome. Patients with creatinine levels ≥2 mg/dL were not eligible.
9. Had use of recreational drugs or history of drug addiction, within the prior 6 months.
10. Had known history of positive hepatitis B surface antigens or hepatitis C virus (HCV) antibodies.
11. Had known history of positive test for human immunodeficiency virus (HIV) antibodies
12. Had psychiatric or neurologic conditions that could have compromised patient safety or compliance, or interfered with the ability to give proper informed consent.
13. Had history of other active malignant disease within 5 years, other than cured basal cell carcinoma of the skin, cured in situ carcinoma of the cervix, or localized prostate cancer that had received definitive therapy. Such prostate cancer patients who were receiving hormonal therapy were eligible.
14. Had the presence of disseminated intravascular coagulation, as confirmed by laboratory studies demonstrating evidence of both increased thrombin generation (decreased fibrinogen, prolonged prothrombin time [PT] and partial thromboplastin time [aPTT]), as well as increased fibrinolysis (elevated D-dimer level).
15. Had received any form of anticoagulant therapy.
16. Had the presence of a known bleeding disorder or coagulation abnormality.
17. Had received treatment with any other investigational agent within 7 days prior to study entry. All prior toxicities should have been resolved to no greater than Grade 1 (with the exception of alopecia).
18. Were pregnant or breast-feeding patients.
19. Were of childbearing potential and were not using adequate contraception.
20. Had any condition that required maintenance of platelet counts at 50,000/μL or higher.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-12; Primary Completion 2015-02 (Actual); Study Completion 2015-06 (Actual)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Greer JP, Baer MR, Kinney MC. Acute Myelogenous Leukemia in Adults. In Wintrobe's Clinical Hematology. Lee GR et al ed. Williams and Wilkins, Baltimore, 2098-2142, 2004.
- [Background] Stroncek DF, Rebulla P. Platelet transfusions. Lancet. 2007 Aug 4;370(9585):427-38. doi: 10.1016/S0140-6736(07)61198-2. PMID 17679020
- [Background] Kuter DJ. What is the potential for thrombopoietic agents in acute leukemia? Best Pract Res Clin Haematol. 2011 Dec;24(4):553-8. doi: 10.1016/j.beha.2011.09.002. Epub 2011 Nov 4. PMID 22127320
- [Background] Trafalis DT, Poulakidas E, Kapsimali V, Tsigris C, Papanicolaou X, Harhalakis N, Nikiforakis E, Mentzikof-Mitsouli C. Platelet production and related pathophysiology in acute myelogenous leukemia at first diagnosis: prognostic implications. Oncol Rep. 2008 Apr;19(4):1021-6. PMID 18357391
- [Background] Stasi R, Bosworth J, Rhodes E, Shannon MS, Willis F, Gordon-Smith EC. Thrombopoietic agents. Blood Rev. 2010 Jul-Sep;24(4-5):179-90. doi: 10.1016/j.blre.2010.04.002. Epub 2010 May 20. PMID 20493600
- [Background] Majka M, Janowska-Wieczorek A, Ratajczak J, Kowalska MA, Vilaire G, Pan ZK, Honczarenko M, Marquez LA, Poncz M, Ratajczak MZ. Stromal-derived factor 1 and thrombopoietin regulate distinct aspects of human megakaryopoiesis. Blood. 2000 Dec 15;96(13):4142-51. PMID 11110685
- [Background] Lambert MP, Rauova L, Bailey M, Sola-Visner MC, Kowalska MA, Poncz M. Platelet factor 4 is a negative autocrine in vivo regulator of megakaryopoiesis: clinical and therapeutic implications. Blood. 2007 Aug 15;110(4):1153-60. doi: 10.1182/blood-2007-01-067116. Epub 2007 May 10. PMID 17495129
- [Background] Lambert MP, Reznikov A, Grubbs A, Nguyen Y, Xiao L, Aplenc R, Rauova L, Poncz M. Platelet factor 4 platelet levels are inversely correlated with steady-state platelet counts and with platelet transfusion needs in pediatric leukemia patients. J Thromb Haemost. 2012 Jul;10(7):1442-6. doi: 10.1111/j.1538-7836.2012.04767.x. No abstract available. PMID 22564375
- [Background] Lambert MP, Xiao L, Nguyen Y, Kowalska MA, Poncz M. The role of platelet factor 4 in radiation-induced thrombocytopenia. Int J Radiat Oncol Biol Phys. 2011 Aug 1;80(5):1533-40. doi: 10.1016/j.ijrobp.2011.03.039. PMID 21740995
- [Background] Joglekar MV, Quintana Diez PM, Marcus S, Qi R, Espinasse B, Wiesner MR, Pempe E, Liu J, Monroe DM, Arepally GM. Disruption of PF4/H multimolecular complex formation with a minimally anticoagulant heparin (ODSH). Thromb Haemost. 2012 Apr;107(4):717-25. doi: 10.1160/TH11-11-0795. Epub 2012 Feb 8. PMID 22318669
- [Background] Lambert MP, Sharma SS, Xiao L, Marcus S et al. 2-O, 3-O-Desulfated Heparin (ODSH) Mitigates Chemotherapy-Induced Thrombocytopenia (CIT) by Blocking the Negative Paracrine Effect of Platelet Factor 4 (PF4) On Megakaryopoiesis. Proceedings of the 54th Annual Meeting of the American Society of Hematology. Abstract 386, 2012.
- [Background] Yang L, Yu Y, Kang R, Yang M, Xie M, Wang Z, Tang D, Zhao M, Liu L, Zhang H, Cao L. Up-regulated autophagy by endogenous high mobility group box-1 promotes chemoresistance in leukemia cells. Leuk Lymphoma. 2012 Feb;53(2):315-22. doi: 10.3109/10428194.2011.616962. Epub 2011 Nov 15. PMID 21864037
- [Background] Kang R, Tang D, Schapiro NE, Livesey KM, Farkas A, Loughran P, Bierhaus A, Lotze MT, Zeh HJ. The receptor for advanced glycation end products (RAGE) sustains autophagy and limits apoptosis, promoting pancreatic tumor cell survival. Cell Death Differ. 2010 Apr;17(4):666-76. doi: 10.1038/cdd.2009.149. Epub 2009 Oct 16. PMID 19834494
- [Background] Rao NV, Argyle B, Xu X, Reynolds PR, Walenga JM, Prechel M, Prestwich GD, MacArthur RB, Walters BB, Hoidal JR, Kennedy TP. Low anticoagulant heparin targets multiple sites of inflammation, suppresses heparin-induced thrombocytopenia, and inhibits interaction of RAGE with its ligands. Am J Physiol Cell Physiol. 2010 Jul;299(1):C97-110. doi: 10.1152/ajpcell.00009.2010. Epub 2010 Apr 7. PMID 20375277
- [Background] Abe R, Shimizu T, Sugawara H, Watanabe H, Nakamura H, Choei H, Sasaki N, Yamagishi S, Takeuchi M, Shimizu H. Regulation of human melanoma growth and metastasis by AGE-AGE receptor interactions. J Invest Dermatol. 2004 Feb;122(2):461-7. doi: 10.1046/j.0022-202X.2004.22218.x. PMID 15009731
- [Background] Logsdon CD, Fuentes MK, Huang EH, Arumugam T. RAGE and RAGE ligands in cancer. Curr Mol Med. 2007 Dec;7(8):777-89. doi: 10.2174/156652407783220697. PMID 18331236
- [Background] Krauel K, Hackbarth C, Furll B, Greinacher A. Heparin-induced thrombocytopenia: in vitro studies on the interaction of dabigatran, rivaroxaban, and low-sulfated heparin, with platelet factor 4 and anti-PF4/heparin antibodies. Blood. 2012 Feb 2;119(5):1248-55. doi: 10.1182/blood-2011-05-353391. Epub 2011 Nov 2. PMID 22049520
- [Background] Von Hoff DD, Ramanathan RK, Borad MJ, Laheru DA, Smith LS, Wood TE, Korn RL, Desai N, Trieu V, Iglesias JL, Zhang H, Soon-Shiong P, Shi T, Rajeshkumar NV, Maitra A, Hidalgo M. Gemcitabine plus nab-paclitaxel is an active regimen in patients with advanced pancreatic cancer: a phase I/II trial. J Clin Oncol. 2011 Dec 1;29(34):4548-54. doi: 10.1200/JCO.2011.36.5742. Epub 2011 Oct 3. PMID 21969517
- [Background] Ellerman JE, Brown CK, de Vera M, Zeh HJ, Billiar T, Rubartelli A, Lotze MT. Masquerader: high mobility group box-1 and cancer. Clin Cancer Res. 2007 May 15;13(10):2836-48. doi: 10.1158/1078-0432.CCR-06-1953. PMID 17504981
- [Background] Sims GP, Rowe DC, Rietdijk ST, Herbst R, Coyle AJ. HMGB1 and RAGE in inflammation and cancer. Annu Rev Immunol. 2010;28:367-88. doi: 10.1146/annurev.immunol.021908.132603. PMID 20192808
- [Background] Takada M, Hirata K, Ajiki T, Suzuki Y, Kuroda Y. Expression of receptor for advanced glycation end products (RAGE) and MMP-9 in human pancreatic cancer cells. Hepatogastroenterology. 2004 Jul-Aug;51(58):928-30. PMID 15239215
- [Background] Taguchi A, Blood DC, del Toro G, Canet A, Lee DC, Qu W, Tanji N, Lu Y, Lalla E, Fu C, Hofmann MA, Kislinger T, Ingram M, Lu A, Tanaka H, Hori O, Ogawa S, Stern DM, Schmidt AM. Blockade of RAGE-amphoterin signalling suppresses tumour growth and metastases. Nature. 2000 May 18;405(6784):354-60. doi: 10.1038/35012626. PMID 10830965
- [Background] Tang D, Kang R, Cheh CW, Livesey KM, Liang X, Schapiro NE, Benschop R, Sparvero LJ, Amoscato AA, Tracey KJ, Zeh HJ, Lotze MT. HMGB1 release and redox regulates autophagy and apoptosis in cancer cells. Oncogene. 2010 Sep 23;29(38):5299-310. doi: 10.1038/onc.2010.261. Epub 2010 Jul 12. PMID 20622903
- [Background] Tang D, Kang R, Livesey KM, Cheh CW, Farkas A, Loughran P, Hoppe G, Bianchi ME, Tracey KJ, Zeh HJ 3rd, Lotze MT. Endogenous HMGB1 regulates autophagy. J Cell Biol. 2010 Sep 6;190(5):881-92. doi: 10.1083/jcb.200911078. PMID 20819940
- [Background] Tang D, Loze MT, Zeh HJ, Kang R. The redox protein HMGB1 regulates cell death and survival in cancer treatment. Autophagy. 2010 Nov;6(8):1181-3. doi: 10.4161/auto.6.8.13367. PMID 20861675
- [Background] Kang R, Tang D, Loze MT, Zeh HJ. Apoptosis to autophagy switch triggered by the MHC class III-encoded receptor for advanced glycation endproducts (RAGE). Autophagy. 2011 Jan;7(1):91-3. doi: 10.1038/cdd.2009.149. Epub 2011 Jan 1. PMID 20978368
- [Background] Cheson BD, Bennett JM, Kopecky KJ, Buchner T, Willman CL, Estey EH, Schiffer CA, Doehner H, Tallman MS, Lister TA, Lo-Coco F, Willemze R, Biondi A, Hiddemann W, Larson RA, Lowenberg B, Sanz MA, Head DR, Ohno R, Bloomfield CD; International Working Group for Diagnosis, Standardization of Response Criteria, Treatment Outcomes, and Reporting Standards for Therapeutic Trials in Acute Myeloid Leukemia. Revised recommendations of the International Working Group for Diagnosis, Standardization of Response Criteria, Treatment Outcomes, and Reporting Standards for Therapeutic Trials in Acute Myeloid Leukemia. J Clin Oncol. 2003 Dec 15;21(24):4642-9. doi: 10.1200/JCO.2003.04.036. PMID 14673054
- [Background] Clopper CJ, Pearson ES. The use of confidence or fiducial limits illustrated in the case of the binomial. Biometrika 26;404-413, 1934.
- [Background] Harrill AH, Roach J, Fier I, Eaddy JS, Kurtz CL, Antoine DJ, Spencer DM, Kishimoto TK, Pisetsky DS, Park BK, Watkins PB. The effects of heparins on the liver: application of mechanistic serum biomarkers in a randomized study in healthy volunteers. Clin Pharmacol Ther. 2012 Aug;92(2):214-20. doi: 10.1038/clpt.2012.40. Epub 2012 Jun 27. PMID 22739141
- [Background] Liu L, Yang M, Kang R, Wang Z, Zhao Y, Yu Y, Xie M, Yin X, Livesey KM, Lotze MT, Tang D, Cao L. HMGB1-induced autophagy promotes chemotherapy resistance in leukemia cells. Leukemia. 2011 Jan;25(1):23-31. doi: 10.1038/leu.2010.225. Epub 2010 Oct 7. PMID 20927132
- [Background] Tang D, Kang R, Zeh HJ 3rd, Lotze MT. High-mobility group box 1 and cancer. Biochim Biophys Acta. 2010 Jan-Feb;1799(1-2):131-40. doi: 10.1016/j.bbagrm.2009.11.014. PMID 20123075

RESULTS

PARTICIPANT FLOW:
Groups:
- Dociparstat: Subjects received the following dosing regimen:
  * Cytarabine (100 mg/m2/day) via continuous intravenous (IV) infusion 24 hours daily for 7 days.
  * Idarubicin (12 mg/m2/day) IV on Days 1, 2, and 3.
  * Dociparstat (4 mg/kg) given over 5 minutes IV, immediately after the idarubicin dose on Day 1, followed by a continuous IV infusion (0.25 mg/kg/hr for 24 hours daily) for a total of 7 days.
Period: Overall Study
Arm/Group | Dociparstat
Started | 12
Completed | 10
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Dociparstat
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: years] — Age collected at site
  years | 54 [21 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Region of Enrollment [Number; unit: participants] — Number of US participants
  participants
    United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Time (Days) to Transfusion-independent Platelet Recovery (Platelet Counts Values ≥ 20,000/μL and ≥ 50,000/μL Without a Platelet Transfusion)
Description: A primary endpoint of this study was evidence of an effect of dociparstat on transfusion independent platelet recovery time. The time (days) to transfusion-independent platelet recovery will be defined as the number of days from the first day of chemotherapy until the first of 5 consecutive days with platelet counts values ≥ 20,000/μL and ≥ 50,000/μL without a platelet transfusion.
Time Frame: Day 1 to Day 35 (35 days)
Population: Count recovery was analyzed after induction on the 10 subjects who received a full induction cycle.
Measure: Mean (Full Range); unit: days
Arm/Group | Dociparstat
Number analyzed (Participants) | 10
days
  Platelet count of ≥20,000/µL | 21.3 [18 to 22]
  Platelet count of ≥50,000/µL | 23.1 [19 to 25]

2. Secondary Outcome: Number of Subjects Who Achieved a Morphologic Complete Remission
Description: A secondary endpoint of this study was to determine whether there was preliminary evidence of an effect of dociparstat on remission rate following cytarabine and idarubicin induction in acute myeloid leukemia (AML) patients, which included complete remission (CR) rate (with neutrophil and platelet count recovery) after the first induction cycle.
  Morphologic CR was defined as absolute neutrophil count (ANC) >1000/μL, platelet count >100,000/μL, <5% bone marrow blasts, no Auer rods, and no evidence of extramedullary disease.
Time Frame: Day 1 to Day 35 (35 days)
Population: All randomized subjects were included in this analysis, including the 2 subjects who did not complete induction.
Measure: Count of Participants; unit: Participants
Arm/Group | Dociparstat
Number analyzed (Participants) | 12
Participants | 11

ADVERSE EVENTS:
Arm/Group | Dociparstat
Serious Adverse Events (participants affected / at risk) | 5/12
Other Adverse Events (participants affected / at risk) | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dociparstat (N=12)
Sepsis (Infections and infestations) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Perirectal abscess (Infections and infestations) | 1 (1)
Acute tubular necrosis (Renal and urinary disorders) | 1 (1)
angioedema (Immune system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No